CLINICAL TRIAL: NCT07053657
Title: The Improvement Effect of Vitamin D on the Cardiovascular Health of Overweight/Obesity Adolescents in China
Brief Title: Effect of Vitamin D on Cardiovascular Metabolic Risk in Overweight/Obesity Adolescents in China
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Yuan Mengyuan, Doctor, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 81250471
Record Dates: First submitted 2025-06-19; First posted 2025-07-08 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-06

CONDITIONS: Cardiometabolic Risk Factors
Keywords: cardiometabolic risk; vitamin D

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Vitamin D3:
  Vitamin D3: 2000 IU per day for 6 weeks (two capsules of 800 IU plus one capsule of 400 IU), followed by 800 IU (one capsule of 800 IU) per day for 6 weeks.
  Interventions: Drug: Dietary Supplement: Vitamin D3
- Placebo Comparator (Placebo Comparator): Vitamin D3 placebo:
  Vitamin D3 placebo (i.e., soybean oil).
  Interventions: Drug: Dietary Supplement: Vitamin D3 placebo

INTERVENTIONS:
Drug: Dietary Supplement: Vitamin D3 — 2000 IU per day for 6 weeks (two capsules of 800 IU plus one capsule of 400 IU), followed by 800 IU (one capsule of 800 IU) per day for 6 weeks.
  Arms: Experimental
Drug: Dietary Supplement: Vitamin D3 placebo — Three capsules for 6 weeks, followed by one capsule for 6 weeks.
  Arms: Placebo Comparator

SUMMARY:
The goal of this randomized controlled clinical trial is to investigate the effects of vitamin D3 supplementation on cardiometabolic risk in Chinese adolescents with overweight/obesity and vitamin D deficiency. The main question it aims to answer whether vitamin D3 supplementation can improve cardiovascular metabolic health.

Participants in the intervention group will receive vitamin D3. The control group will receive vitamin D placebo.

Researchers will compare the change in cardiometabolic risk from baseline to post-intervention at 12 weeks between the intervention and control groups.

DETAILED DESCRIPTION:
Investigators will conduct a randomized controlled trial to examine whether vitamin D3 supplementation can improve cardiovascular metabolic health. A total of 130 participants will be recruited from two middle schools. Inclusion criteria were students with both students and parents signing a paper version of the informed consent form, overweight/obesity and serum 25(OH)D concentration of 12~20ng/ml. Exclusion criteria are any disease that affects vitamin D metabolism (e.g., functional/organic brain disease, severe infectious disease, chronic gastrointestinal disease, hepatic or renal insufficiency, etc.); known chronic disease (e.g., cardiovascular disease); use of vitamin D supplements in the past 3 months; and adolescents with allergies to vitamin D or soybean oil ingredients. Participants will be randomly assigned into a supplementation or placebo group. Supplementation arm will receive oral dose 2000 IU vitamin D3 per day for 6 weeks and followed by 800 IU per day for 6 weeks, placebo arm will receive placebo every day for 12 weeks. For the first 6 weeks, vitamin D or placebo will be administrated every two weeks. For the next 6 weeks, vitamin D or placebo will be administrated every 3 weeks. The primary outcome of this study is to compare the change of cardiometabolic risk between supplementation or placebo group from post-intervention 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Students whose caregivers signed informed consents;
2. Students with serum 25(OH)D concentration of 12-20 ng/mL;
3. Students with overweight or obesity.

Exclusion Criteria:

1. Students with any disease that affects vitamin D metabolism (e.g., functional/organic brain disease, severe infectious disease, chronic gastrointestinal disease, hepatic or renal insufficiency, etc.);
2. Students with known chronic disease (e.g., cardiovascular disease); use of vitamin D supplements in the past 3 months;
3. Students with allergies to vitamin D or soybean oil ingredients.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in cardiometabolic risk scores | From randomization to the end of intervention at 3 months
  The cardiovascular metabolic risk scores was the sum of the sex-specific standardized z-score for 5 indicators: WC, MAP (MAP=1/3*SBP+2/3*DBP), HDL-C (HDL-C value multiplied by -1), TG, and fasting glucose. A higher cardiometabolic risk scores indicates a higher individual cardiometabolic risk. Change in cardiometabolic risk scores from pre to post-intervention were compared between randomized groups, which was the primary outcome of this study

SECONDARY OUTCOMES:
BMI | From randomization to the end of intervention at 3 months
  Measurements were taken by trained researchers using a height and weight meter. The instrument was calibrated before the measurement and the subjects were asked to remove their shoes and wear light clothes during the measurement. We used weight in kilograms and height in metres to calculate BMI. The unit of BMI is kg/m^2, BMI=Weight/(Height*2) in kg/m^2.
Waist circumference and Sum of skinfold thickness | From randomization to the end of intervention at 3 months
  Subcutaneous fat thickness was measured in the upper arm (at the midpoint of the line between the acromion point and the ulnar humerus), subscapularis (1 cm below the subscapularis) and abdomen (junction of the right midclavicular line and the umbilical level) using a skinfold thickness gauge after uniform training, with the results expressed in mm to one decimal place, and all of which required zeroing and pressure testing work of the skinfold thickness gauge before use. Waist circumference was measured using a corrected tape measure, circling horizontally along the midpoints of the lower edge of the ribs and the upper edge of the hip bone, and readings were recorded at the end of expiration to an accuracy of 0.1 cm.
Blood pressure | From randomization to the end of intervention at 3 months
  The researchers measured systolic and diastolic blood pressure using an Omron HEM-7124 digital sphygmomanometer. Measurements were taken with the subject in a sitting position and started after 10 minutes of sitting still, with 2 measurements taken at 5 minute intervals. The average of the two measurements will be taken.
Blood glucose and lipid | From randomization to the end of intervention at 3 months
  After each subject fasted overnight, the next day two professional nurses took their fasting blood samples by venipuncture, the blood samples were stored in an insulated box with ice packs, and all the samples were immediately transported to the laboratory to be tested by the professionals, and the indexes measured included fasting blood glucose, total cholesterol, triglycerides, HDL cholesterol and LDL cholesterol.
TyG index | From randomization to the end of intervention at 3 months
  TyG index is considered an important predictor of IR risk and can be used to screen children and adolescents to prevent cardiovascular disease in adulthood. TyG index=ln (Triglyceride * Fasting bolld glucose) - ln (2).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Anhui Medical University, Anqing, Anhui
  - Anhui Medical University, Hefei, Anhui

IPD SHARING:
Plan to Share IPD: No
IPD will be only used in a peer-reviewed journal in order to protect the privacy of the study participants.